CLINICAL TRIAL: NCT00211133
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Impact of Maintaining Hemoglobin Using Eprex (Epoetin Alfa) in Metastatic Breast Carcinoma Subjects Receiving Chemotherapy
Brief Title: A Study to Evaluate the Impact of Maintaining Hemoglobin Levels Using Epoetin Alfa in Patients With Metastatic Breast Cancer Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004414
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Anemia; Breast Neoplasms; Quality of Life
Keywords: Anemia; Breast Cancer; Breast Tumor; Quality of Life; Women; Female; Chemotherapy; Hemoglobin; Survival; Epoetin; Epoetin alfa; erythropoietin
MeSH Terms: conditions — Anemia; Breast Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the impact on survival and quality of life of maintaining hemoglobin in the range of 12 to 14 g/dL using epoetin alfa or placebo in patients starting chemotherapy for metastatic breast cancer for the first time.

DETAILED DESCRIPTION:
Cancer patients often experience anemia due to the disease itself, chemotherapy or both. Quality of life is also affected, due in part to the fatigue associated with anemia. Previous studies with epoetin alfa have suggested that achieving a higher hemoglobin level may improve quality of life and help patients live longer.This randomized, double-blind, placebo-controlled multi-center study evaluated the effects of treatment with epoetin alfa in maintaining hemoglobin levels between 12 and 14 g/dL to determine its impact on survival and quality of life, in addition to investigating the possible role that epoetin alfa may have on tumor response to chemotherapy. During the double-blind portion of the study, patients were to receive 12 months of treatment with epoetin alfa or placebo. Thereafter, follow-up evaluations were to occur every 3 months until 75% of the patients had died. Effectiveness was to be determined by recording the number of patients surviving at 12 months, the change in hemoglobin from the start of the study until study completion, response to chemotherapy and quality of life. Safety evaluations (incidence of adverse events, physical examinations and clinical laboratory tests) were to be performed throughout the study. The study hypothesis was that maintaining hemoglobin in the range of 12 to 14 g/dL would improve 12-month survival and quality of life in patients with metastatic breast cancer who were receiving chemotherapy. Since the time this study was originally designed, the prescribing information for epoetin alfa has changed. Current use of epoetin alfa should follow the prescribing information. Patients were to receive epoetin alfa injections (40,000 units) under their skin once per week for 12 months or matching placebo. Dosage was to be adjusted up (to 60,000 units) or down (to 75% of the last dose administered) as needed to maintain hemoglobin levels between 12 and 14 g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Female patients >= 18 years of age with confirmed diagnosis of metastatic breast cancer who are predicted to start chemotherapy for the first time
* Weight > = 40 kg (88 lbs)
* Postmenopausal for at least 1 year, surgically sterile or practicing an effective method of birth control and have a negative serum pregnancy test at the start of the study
* Must have signed an informed consent

Exclusion Criteria:

* Clinically significant lung, heart, hormone, neurological, gastrointestinal, urinary tract or reproductive system disease
* Receiving dose intensification chemotherapy for bone marrow or stem cell transplantation
* Cancer of the brain or brain/spinal cord disease
* Locally advanced or inflammatory breast cancer as the only symptom of breast cancer
* Active second primary cancer or documented history of other cancer within the last 3 years
* Anemia from a cause other than cancer or radiotherapy/chemotherapy
* History of stoke, clots in the lungs or legs or any other blood clotting disorders
* Uncontrolled high blood pressure
* Untreated folate or Vitamin B12 deficiency
* Treatment with epoetin alfa or other forms of erythropoietin within the last 4 weeks
* Known hypersensitivity to epoetin alfa or any of its components
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2000-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
12-month survival rate, defined as the proportion of patients alive at 12 months after the start of the study.

SECONDARY OUTCOMES:
Hemoglobin and change in hemoglobin. End of chemotherapy/end of study tumor response. Quality of life. Overall 12-month survival. Red blood cell transfusion rates. Time-to-cancer progression. Overall/median survival times.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Leyland-Jones B, Semiglazov V, Pawlicki M, Pienkowski T, Tjulandin S, Manikhas G, Makhson A, Roth A, Dodwell D, Baselga J, Biakhov M, Valuckas K, Voznyi E, Liu X, Vercammen E. Maintaining normal hemoglobin levels with epoetin alfa in mainly nonanemic patients with metastatic breast cancer receiving first-line chemotherapy: a survival study. J Clin Oncol. 2005 Sep 1;23(25):5960-72. doi: 10.1200/JCO.2005.06.150. Epub 2005 Aug 8. PMID 16087945